CLINICAL TRIAL: NCT03849976
Title: Evaluation of the Impact of the Therapeutic Communication Training of the Stretcher Bearers on the Patient Anxiety in the Operating Room (STRESSCOM)
Brief Title: Therapeutic Communication Training of the Stretcher Bearers on the Patient Anxiety (STRESSCOM)
Acronym: STRESSCOM
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0075
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Anxiety
Keywords: Therapeutic communication; Anxiety; Endoscopic examination under general anesthesia; Operating room; Stretcher bearer
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Patients accompanied to the operating room by a stretcher bearer trained in therapeutic communication
  Interventions: Behavioral: Therapeutic communication
- Control group: Patients accompanied to the operating room by a stretcher bearer not trained in therapeutic communication

INTERVENTIONS:
Behavioral: Therapeutic communication — Patients will be accompanied to the operating room by a stretcher bearer trained in therapeutic communication
  Groups: Experimental group

SUMMARY:
Anxiety is a form of psychic and/or physical discomfort caused by the feeling of the imminence of a danger. It is a frequent perioperative manifestation of patients. Pharmacological premedication is currently used to avoid perioperative anxiety. However, its effect is now controversial and non-drug techniques have been also studied.

The therapeutic communication aims to provide analgesia or anxiolysis to enhance the patient's well-being and to separate the patient from the surrounding reality through the suggestion of positive images with a chosen verbal and nonverbal approach. This prospective, monocentric, comparative, double-blind study aims to evaluate the impact of the training of stretcher-bearers in therapeutic communication on the anxiety of patients who go to the operating room for an endoscopic examination under general anaesthesia.Two groups of patients will be compared: In the first group patients will be accompanied to the operating room by a stretcher-bearer trained in therapeutic communication, in the second group patients will be accompanied by a stretcher bearer without this specific training.

DETAILED DESCRIPTION:
Anxiety is a form of psychic and/or physical discomfort caused by the feeling of the imminence of a danger. It is a normal reaction of adaptation and defense face to a situation lived as hostile. It is a frequent perioperative manifestation. Patients who need an intervention are indeed 20% more anxious than the general population. The occurrence of this anxiety can have consequences for perioperative medical care influencing morbidity and mortality.

Pharmacological premedication initially prescribed in the 19th century to limit the adverse effects of general anesthesia is currently used to fight perioperative anxiety. However, its effects are now considered as controversial.

and non-drug techniques have been studied. They have the advantage of being inexpensive and causing little or no adverse effects.

Therapeutic communication can be defined as a relational technique that seeks to separate the patient from the surrounding reality to provide analgesia or anxiolysis through the suggestion of positive images with a chosen verbal and nonverbal approach.

The knowledge of communication techniques resulting from hypnosis by the healthcare team could therefore optimize patient medical care in terms of analgesia and the management of perioperative anxiety. Therapeutic communication training in the operating room is short and accessible to all members of the team regardless of their rank. This is a training provided internally by a certified practitioner in therapeutic hypnosis, aiming to give to the professionals knowledge to optimize the patient support. At the hospital (Groupement des Hôpitaux de l'Institut Catholique de Lille), several stretcher bearers have been trained in therapeutic communication and are already applying it routinely.

No study has yet investigated the impact of the use of therapeutic communication in the operating room to control the level of anxiety of patients.

This study is prospective, monocentric, comparative, double blind. Two groups of patients will be compared: In the first group patients will be accompanied to the operating room by a stretcher-bearer trained in therapeutic communication, in the second group patients will be accompanied by a stretcher bearer without this specific training.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Hospitalized in the ambulatory sector for endoscopic examination under general anesthesia (fibroscopy/colonoscopy/others)
* Able to answer anxiety questionnaires
* Able to walk to the operating room according to the usual practice (no motor disorder)
* Not presenting a psychiatric or cognitive disorder, or a non-paired hearing disorder that may interfere with therapeutic communication
* Being informed and not being opposed

Exclusion Criteria:

* Refusal to participate in the study
* Patients under guardianship
* Patient who received premedication before going down to the operating room (benzodiazepines, gabapentin, antihistamines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in ambulatory sector for endoscopic examination under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Anxiety scale: State-Trait Anxiety Inventory (STAI-Y), form A | Day one (before intervention)
  This scale is composed of 20 propositions to know how the subject feels. Each item has a score from 1 to 4 (4 being the highest degree of anxiety). The score therefore varies from 20 to 80.
Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Day one (before intervention)
  The APAIS questionnaire includes 6 questions, 2 of which evaluate the patient's anxiety about anesthesia, 2 questions estimate the anxiety about the procedure, the last 2 questions evaluate the patient's need for information about anesthesia and the procedure. Each question is rated from 1 to 5, the scale allows to calculate 4 scores (anesthetic anxiety/intervention anxiety/global and information request score). Subjects are considered anxious when they have a score higher than 11 for these 4 items.

SECONDARY OUTCOMES:
Evaluation of the experience of general anesthesia (EVAN-G) scale | In average one day (at hospital discharge)
  EVAN-G questionnaire includes 26 questions. Results are grouped together to define 6 "dimensions": Focus of attention, Information, Privacy, Pain, Discomfort and Waiting Times. From these scores, an overall satisfaction score is calculated (average of all scores). For each of the scores: the higher the score, the higher the satisfaction.
Likert scale | Day one (at the end of the intervention)
  Patient cooperation: evaluated by the nurse anesthesiologist with a Likert scale rated from 1 (no cooperation) to 5 (excellent cooperation).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Canevet, Principal Investigator — Lille Catholic University
Locations (1):
- Lille Catholic Hospitals, Lomme, Nord, France

IPD SHARING:
Plan to Share IPD: No